CLINICAL TRIAL: NCT00225550
Title: Dose Finding, Safety, Pharmacokinetic and Pharmacodynamic Study of the Vascular Targeting Agent Exherin™ (ADH-1) Administered Once Daily for 5 Consecutive Days by Intravenous Infusion in Subjects With N-Cadherin Expressing, Incurable, Solid Tumors (Adherex Protocol Number AHX 01 003)
Brief Title: A Study of the Safety and Effects of ADH-1 Given Daily to Subjects With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adherex Protocol AHX-01-003
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2007-08-06 (Estimated); Status verified 2007-08

CONDITIONS: Neoplasms
Keywords: Cancer;; Tumors;; Neoplasms;; Anticarcinogenic Agents;; Antineoplastic Agents;; Cadherins
MeSH Terms: conditions — Neoplasms | interventions — N-Ac-CHAVC-NH2

INTERVENTIONS:
Drug: ADH -1 (Exherin™)

SUMMARY:
N-cadherin, a protein involved in blood vessel cell binding, is increased as cancer progresses, and is on the surface of many tumor cells. ADH-1 blocks N-cadherin. This study will test the safety and effects of ADH-1 in subjects with incurable, solid tumors with a protein biomarker called N-cadherin. This study will identify the amount of ADH-1 that subjects can tolerate.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Male and female patients > or = 18 years of age with a solid tumor(s) refractory to standard curative therapy or for which no curative therapy exists
* Clinically or radiologically documented measurable disease.
* Immunohistochemical evidence of N-cadherin expression (at least 1+ positive) in archived or fresh tumor tissue
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing and electrocardiogram (ECG)

Exclusion criteria:

* Receipt of ADH-1 prior to this clinical study
* Chemotherapy, radiotherapy, or any other investigational drug within 30 days before study entry
* History of primary brain tumors or brain metastases
* History of spinal cord compression or tumors that have shown any evidence of active bleeding within 30 days before study entry.
* Stroke, major surgery, or other major tissue injury within 30 days before study entry
* History of congestive heart failure, myocardial infarction, angina, life threatening arrhythmias, significant electrocardiogram (ECG) abnormalities, or known hypercoagulable states

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com